CLINICAL TRIAL: NCT06003192
Title: Screen Smart: Using Digital Health to Improve HIV Screening and Prevention for Adolescents in the Emergency Department
Brief Title: Screen Smart: Using Digital Health to Improve HIV Screening and Prevention
Acronym: Screen Smart
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1R01HD110321-01A1 (NIH)
Record Dates: First submitted 2023-08-03; First posted 2023-08-21 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-02

CONDITIONS: HIV Infections
Keywords: HIV; adolescents; emergency department; mHealth; preventive care
MeSH Terms: conditions — HIV Infections; Emergencies

STUDY DESIGN:
Intervention Model Description: Interrupted Times Series Model
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Universal Opt-out HIV Screening (Other): The intervention is offering universal opt-out HIV screening to all adolescents 15 to 21 years of age that are seeking care in the emergency department.
  Interventions: Other: Universal Opt-out HIV Screening

INTERVENTIONS:
Other: Universal Opt-out HIV Screening — Using a tablet device, offering universal opt-out HIV screening to adolescents seeking care in a pediatric emergency department.

SUMMARY:
The goal of this interrupted time series quasi-experimental design study is to implement universal opt- out HIV testing and linkage to HIV preventive care in 15-21 year old adolescents visiting the pediatric emergency department (ED). The main question[s] it aims to answer are:

1. What is the uptake, reach and effectiveness of universally offered, opt-out HIV screening across pediatric EDs after implementing an adapted version of a tablet-based screening process?
2. What is the successful linkage to comprehensive HIV pre-exposure prophylaxis (PrEP) care using a novel, digital health platform? Participants will

   1. Complete the previously developed and validated computerized sexual health screen (cSHS) containing questions regarding their personal sexual health history
   2. Have the opportunity to opt-out of clinician-ordered HIV testing
   3. Patients meeting CDC criteria for HIV PrEP will be given the opportunity to enroll in the digital health PrEP linkage platform and followed for 3 months after enrollment.

DETAILED DESCRIPTION:
Using a previously developed tablet-based, broad scale gonorrhea and chlamydia screening process, the investigators will adapt, refine, and test this process with the aim of increasing universally offered, opt-out HIV screening in the pediatric ED through electronic integration of patient reported data for provision of clinical decision support for HIV screening and identification of PrEP candidacy. The investigators will then use mHealth to link patients to PrEP services. The goal of this study is to (1) adapt, refine, and test this previously implemented multi-center, ED-based, screening study with a goal of increasing universally offered, opt-out HIV screening among adolescents in the pediatric ED and (2) link at-risk adolescents to PrEP services and preventive care. This will be accomplished through a network of children's hospital EDs (Pediatric Emergency Care Applied Research Network or PECARN). This research will contribute to the evidence base for creating clinically effective and sustainable HIV screening programs that can be successfully implemented into the clinical workflow of the ED. It will also improve identification and linkage to PrEP care for at risk adolescents using mHealth strategies by first identifying adolescents and young adults (AYA) who are PrEP candidates based on their responses to a computerized sexual health screen (cSHS) and subsequently (1) providing clinical decision support to providers via the electronic health record and (2) direct text messaging from the cSHS to PrEP candidates providing educational content and connecting youth to a PrEP navigator. This intervention will rely on an innovative approach that electronically integrates patient-reported data to guide clinical decision support.

ELIGIBILITY:
Inclusion Criteria:

* All patients 15-21 years of age visiting a pediatric emergency department.

Exclusion Criteria:

* Unable to understand English
* Critically ill
* Cognitively impaired
* Altered mental status

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 63000 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
HIV testing rates per 1000 eligible patients during each month | 30 months
  We will employ interrupted time series analyses to compare these rates between baseline (usual care) and upon implementation of universally offered, opt-out HIV screening strategy.
HIV infection rates per 1000 eligible patients during each month | 30 months
  We will employ interrupted time series analyses to compare these rates between baseline (usual care) and upon implementation of universally offered, opt-out HIV screening strategy
Linkage of PrEP | 30 months
  The number of PrEP eligible youth who are enrolled in the mHealth platform and complete a followup appointment in their comprehensive PrEP care medical home within 1 month of the ED visit.

SECONDARY OUTCOMES:
Identification of PrEP eligible and interest in starting PrEP | 30 months
  The proportion of patients who are identified as PrEP eligible and who endorse interest in starting PrEP
Demographics associated with PrEP eligibility | 30 months
  Sociodemographic and visit characteristics associated with PrEP eligibility.
Demographics associated with PrEP linkage to care | 30 months
  Sociodemographic and visit characteristics associated with completion of PrEP care visit within 1 month of study enrollment.
Demographics associated with HIV screening acceptance | 30 months
  Sociodemographic and visit characteristics associated with patient HIV screening acceptance
HIV positivity rates in different sexual risk strata | 30 months
  Comparison of HIV positivity rates between patients in the different sexual risk strata (determined by patient entered cSHS)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Reed, MD, MS, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Monika Goyal, MD, MSCE, Principal Investigator — Children's National Research Institute; Nadia Dowshen, MD, MSHP, Principal Investigator — Children's Hospital of Philadelphia
Locations (4):
- United States (4):
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - Children's Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No